CLINICAL TRIAL: NCT00649831
Title: Azithromycin (Zithromax®) 5 Days Versus Amoxicillin-Clavulanic Acid (Augmentin®): Multicentre, Randomised, Open-Label Study To Compare The Clinical Efficacy And Safety Of Azithromycin With Those Of Amoxicillin-Clavulanic Acid In Patients Presenting With An Exacerbation Of Chronic Bronchitis
Brief Title: A Multicentre, Randomised, Open-Label Study To Compare The Efficacy And Safety Of Azithromycin For 5 Days With Those Of Amoxicillin-Clavulanic Acid In Patients With Chronic Bronchitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0661045
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Bronchitis, Chronic
MeSH Terms: conditions — Bronchitis, Chronic | interventions — Amoxicillin; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2 (Active Comparator)
  Interventions: Drug: Amoxicillin/clavulinic acid
- Group 1 (Active Comparator)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Amoxicillin/clavulinic acid — amoxicillin/clavulinic acid 500 mg/62.5 mg tablet; take 2 tablets by mouth twice daily (BID) for 10 days
  Arms: Group 2
Drug: Azithromycin — Azithromycin 250 mg tablet; take 2 tablets by mouth on the first day, then 1 tablet by mouth from Days 2 to 5
  Arms: Group 1

SUMMARY:
This study compared the clinical efficacy and safety of azithromycin with that of amoxicillin-clavulanic acid, in patients between the ages of 35 and 75 years, presenting with an exacerbation of chronic bronchitis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Outpatients presenting with an exacerbation of chronic bronchitis including: chronic bronchitis with obstructive respiratory disorders documented by a forced expiratory volume of below 80% and higher than 35% of the theoretical value, within the previous 12 months; and thought to be of infectious origin

Exclusion Criteria:

Exclusion Criteria:

* Patient not presenting with the associated signs of an exacerbation
* Patient presenting with clinical signs suggestive of pneumonopathy at inclusion
* Patient requiring hospitalisation in intensive care

Ages: 36 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2002-10; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
To assess clinical efficacy (clinical recovery or clinical failure) | Day 30

SECONDARY OUTCOMES:
Number of exacerbations | Day 30 to Day 90
Bacteriological monitoring (a descriptive analysis of streptococci in the bacterial flora and their sensitivity to antibiotics at the different collections of sputum) | continuous

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- France (27):
  - Pfizer Investigational Site, Anzin
  - Pfizer Investigational Site, Avignon
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Escaudain
  - Pfizer Investigational Site, Équeurdreville-Hainneville
  - Pfizer Investigational Site, Le Grand-Quevilly
  - Pfizer Investigational Site, Les Lilas
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Mantes-la-Jolie
  - Pfizer Investigational Site, Maromme
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Maubeuge
  - Pfizer Investigational Site, Mont-Saint-Martin
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Saint-Aulaire
  - Pfizer Investigational Site, Savigny
  - Pfizer Investigational Site, Soissons
  - Pfizer Investigational Site, Tourcoing
  - Pfizer Investigational Site, Tulette
  - Pfizer Investigational Site, Valenton
  - Pfizer Investigational Site, VAUX S/ Seine
  - Pfizer Investigational Site, Villejuif
  - Pfizer Investigational Site, Vincennes
  - Pfizer Investigational Site, Vitry
  - Pfizer Investigational Site, Wattrelos
  - Pfizer Investigational Site, Yerres

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661045&StudyName=A%20Multicentre%2C%20Randomised%2C%20Open-Label%20Study%20To%20Compare%20The%20Efficacy%20And%20Safety%20Of%20Azithromycin%20For%205%20Days%20With%20Those%20Of%20Amoxicillin-